CLINICAL TRIAL: NCT04966494
Title: Effect of the Consumption of a Common Bean (Phaseolus Vulgaris L.) and Oats Snack Bar on the Proteomic Profile of Human Mononuclear Cells
Brief Title: Impact of Beans and Oats Snack Bar on Hypertriglyceridemic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Responsible Party: Principal Investigator, Ivan Luzardo-Ocampo, Associate Researcher, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20131004
Record Dates: First submitted 2021-07-02; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Hypertriglyceridemia; Obesity
Keywords: Common beans; Oats; Proteomic Analysis; Phenolic compounds; Dietary Fiber
MeSH Terms: conditions — Hypertriglyceridemia; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOSB Group (Experimental): This group consumed a common beans and oats snack bar (BOSB) for 8 weeks.
  Interventions: Dietary Supplement: BOSB
- Control Group (No Intervention): This group corresponded to hypertriglyceridemic women who does not consume BOSB

INTERVENTIONS:
Dietary Supplement: BOSB — BOSB consisted on a oats (26 %), common beans (30 %), water and emulsifier-based snack bar, administered daily (50 g/day) during 8 weeks.
  Arms: BOSB Group

SUMMARY:
Hypertriglyceridemia is a serious condition in the Mexican population and it is considered a major risk factor for cardiovascular disease. Current efforts to prevent dyslipidemia and lipids alteration include the development of functional products as an alternative for the management of hypertriglyceridemia. Common beans (Phaseolus vulgaris L.) are a recognized good source of bioactive compounds, mainly phenolic compounds, total dietary fiber (insoluble and soluble fiber, resistant starch and oligosaccharides), saponins, and phytosterols that exert hypolipidemic effects. In this sense, the development of beans-based food products is an alternative for improving the general health status. In previous work, a beans-oats snack bar formulation was found to be a promising potential functional product. In order to validate those results, the aim of this works was to assess a clinical trial was conducted with Mexican women to assess the effect of daily consumption of the functional product on serum triglycerides and certain plasma proteins involved in lipids metabolism in a clinical trial. The clinical trial was 2 months, randomized parallel study where 32 women with elevated triglycerides were randomized into the treatment group and control group. The Control group received nutritional orientation whereas the treatment group received the orientation and consumed 50 g of the product per day. Fasting blood samples were collected at baseline and the end of the study, obtaining serum and plasma for analysis of lipids profile, glucose, and biomarkers. To determine changes in plasma proteins, a 182 protein Human Obesity Antibody Array was used, and the results were analyzed using a bioinformatic-based analysis from Ingenuity Pathways Analysis (QIAGEN)

ELIGIBILITY:
Inclusion Criteria:

* No current diagnoses of illnesses.
* Triglycerides levels among 150 and 350 mg/dL.
* No allergies to common beans and oats.
* Not pregnant or lactating.

Exclusion Criteria:

* If they had current diagnoses of diabetes, hypertension, irritable bowel syndrome, or cancer.
* Taking anti-inflammatory drugs.
* Fasting glucose >100 mg/dL, total cholesterol >240 mg/dL, LDL C>160 mg/dL.
* Reported intolerances to BOSB ingredients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10-05 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2015-11-02 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 8 weeks
  Significant change
Glucose | 8 weeks
  Significant change

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Loarca-Piña, Ph. D., Principal Investigator — Universidad Autonoma de Queretaro

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: ICF, CSR
Time Frame: 10 years

REFERENCES:
- [Derived] Ramirez-Jimenez AK, Luzardo-Ocampo I, Cuellar-Nunez ML, Anaya-Loyola MA, Leon-Galvan MF, Loarca-Pina G. Daily Intake of a Phaseolus vulgaris L. Snack Bar Attenuates Hypertriglyceridemia and Improves Lipid Metabolism-Associated Plasma Proteins in Mexican Women: A Randomized Clinical Trial. Front Nutr. 2022 Jun 3;9:890136. doi: 10.3389/fnut.2022.890136. eCollection 2022. PMID 35719139